CLINICAL TRIAL: NCT01001780
Title: Pentostatin, Cyclophosphamide Plus Rituximab (PCR) for the Therapy of Poor-Prognosis Chronic Graft-Versus-Host Disease
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study stopped early due to poor accrual.
Sponsor: University of Rochester (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25260
Record Dates: First submitted 2009-10-26; First posted 2009-10-27 (Estimated); Last update posted 2013-10-16 (Estimated); Status verified 2013-10

CONDITIONS: Active Chronic Graft Versus Host Disease
Keywords: Graft versus Host Disease; Allogeneic Hematopoietic Stem Cell Transplant
MeSH Terms: conditions — Graft vs Host Disease | interventions — Pentostatin; Cyclophosphamide; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pentostatin, Cyclophosphamide, Rituximab (Experimental)
  Interventions: Drug: Pentostatin; Cyclophosphamide; Rituximab

INTERVENTIONS:
Drug: Pentostatin; Cyclophosphamide; Rituximab — Pentostatin 2mg/m2 IV day+1 (up to 6 cycles) Cyclophosphamide 600mg/m2 IV day+1 (up to 6 cycles) Rituximab 375mg/m2 IV day+1 (up to 6 cycles)
  Other Names: Pentostatin - Nipent; Cyclophosphamide - Cytoxan; Rituximab - Rituxan

SUMMARY:
Chronic graft-versus-host disease (GvHD) is a severe, life threatening complication from getting a bone marrow or stem cell transplant. It is caused by certain cells from the donor that attack your cells. The usual treatments, prednisone and cyclosporine, don't work very well in chronic GVHD.

This research is being done to determine if the combination of the chemotherapeutic and immunosuppressive, drugs pentostatin, cyclophosphamide and the monoclonal antibody rituximab, used as in the "PCR" combination will prove useful in the treatment of certain patients with chronic GvHD (namely those who are unlikely to respond to standard therapy).

DETAILED DESCRIPTION:
As above, your chronic GvHD either has not responded to, or is not expected to, respond to standard immunosuppressive treatment for chronic GvHD. These standard treatments are given in relatively low doses over long intervals. Thus, in this study we are testing an alternate strategy, using a more intensive, combined therapy with the PCR combination to determine if it will improve outcomes. PENTOSTATIN, CYCLOPHOSPHAMIDE plus RITUXIMAB ("PCR") are FDA-approved drugs for chemotherapy of certain lymphomas/leukemias, and although each has been used separately to treat patients with chronic GvHD, they have not been approved as immunosuppressant for the treatment of chronic GvHD, either separately or together. We will study the "PCR" combination in 9-17 patients with chronic GvHD who are refractory to, or not expected to respond to standard therapy. Response will be measured by the achievement of a documented complete remission (i.e., full resolution of all symptoms and signs), and thus, a shortening of the total duration of immunosuppressive (anti-chronic GvHD) therapy. This latter effect may reduce overall infections.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic GvHD requires at least one diagnostic and/or at least one distinctive manifestation. The latter must be confirmed by pertinent biopsy, laboratory tests, or radiology in the same or another organ. (See 19.11 details)
* Confirmation of active chronic GvHD is desired but may not be feasible.
* Age >/= 18 yrs. No gender or ethnic restrictions.
* Previously untreated chronic GvHD
* Up to 15 days' of single agent therapy may be given for patients to be considered "previously-untreated", provided progression is not observed.
* Vogelsang score20 >/= 2
* If patients progress while on prednisone >/= 0.5 mg/kg/day (or equivalent) for treatment of acute GvHD as they develop chronic GvHD, they may be considered candidates irrespective of the Vogelsang Score.
* Prior therapy. Patients must have received prednisone >/= 0.5 mg/kg/day plus one (or more) of the following second agents: tacrolimus, cyclosporine, sirolimus, or mycophenolate.
* All second and subsequent failures are eligible.
* Special circumstances: involvement of a "critical organ". In these cases, progressive involvement after the use of initial therapy will suffice as a eligibility criteria irrespective of the Vogelsang score.

Exclusion Criteria:

* Previous history of severe adverse reaction to either study agent.
* Prior exposure alone to any of the agents in PCR is not a contraindication, Use of more than one of the agents in PCR to treat GvHD will exclude patients from entry.
* Serious active infection (especially hepatitis B or C) not responding to therapy.
* Active malignancy and/or the requirement of immunomodulation as treatment of malignancy.
* Hematologic abnormalities: WBC <3.0 K/uL, ANC < 1.0 K/uL, Hgb < 8.0 g/dL, platelets < 50.0 K/uL.
* Non-hematologic toxicities*:
* *Renal. Measured creatinine clearance <35 ml/min or the concomitant need for dialysis.
* *Pulmonary. DLCO <40%, FEV1, 50%.
* *Hepatic. LFT (as measured by AST, ALT, T.bili) One or all of the levels found to be >3 x normal.
* Other. History of any significant co-morbid disease felt to make proposed therapy excessively risky.
* Psychiatric. Patients with uncompensated severe psychiatric illness that would preclude signing the necessary consent forms or being compliant.
* Compliance. Patients unlikely to adhere to study procedure and/or is unable or unwilling to return for necessary follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-08; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Determine whether complete response rate following use of PCR regimen exceeds 25% in selected (for poor prognosis) chronic GvHD patients. | One year
Assess the ability to successfully wean patients from all immunosuppressive therapy following complete response. | One year

SECONDARY OUTCOMES:
Describe the incidence, frequency and type of all observed opportunistic infections. | One year
Describe the pattern of immune recovery in these patients | One year
Assess the incidence, frequency and type of hematologic dysfunction before and after therapy. | One year
Assess the incidence of relapse (of the underlying malignant diagnosis for which the allogeneic hematopoietic stem cell transplant was performed), progression-free and overall survival. | One year

CONTACTS AND LOCATIONS:
Overall Officials: Gordon Phillips, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States